CLINICAL TRIAL: NCT03114579
Title: Evaluation of the Measurement of Cardiac Output by the NEXFIN HD Monitor in Peroperative
Acronym: NEXFIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0005
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Output; Peroperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measure of the cardiac output obtained by a reference methode (Other)
  Interventions: Device: Intraoperative heart rate measurement (reference method)
- Measurement of cardiac output obtained by NEXFIN HD. (Other)
  Interventions: Device: NEXFIN HD

INTERVENTIONS:
Device: Intraoperative heart rate measurement (reference method) — Measurement of cardiac output by both monitors: NEXFIN HD and oesophageal doppler, blood pressure measurement by the catheter and NEXFIN HD monitor, and cardiac output and blood pressure measurements after treatment administration (vasoconstrictor or filling)
  Arms: Measure of the cardiac output obtained by a reference methode
Device: NEXFIN HD
  Arms: Measurement of cardiac output obtained by NEXFIN HD.

SUMMARY:
Continuous perioperative cardiac output (DC) and blood pressure (PA) monitoring contributes to hemodynamic stability and ensures adequate perfusion pressure, resulting in a reduction in morbidity and mortality and length of hospital stay.

The monitors usually used in perioperative are either semi-invasive and difficult for calibration (oesophageal Doppler) or invasive (arterial catheter).

The Nexfin HD allows these two measurements and it is completely non-invasive, remains to validate its use in peroperative.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients candidate for surgery under general anesthesia requiring oesophageal Doppler or arterial catheter hemodynamic monitoring.

Exclusion Criteria:

* Patients with cardiac and thoracic surgery,
* patients for whom access to the head is impossible,
* facial trauma patients,
* patients with aortic malformation, dilation or coarctation,
* patients with aortic dissection,
* patients with vascular surgery with aortic clamping,
* patients with a tumor, stenosis or varices of the esophagus,
* patients with severe oesophagitis,
* patients with thoracic radiotherapy
* patients under guardianship or curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2017-02-11 (Actual)

PRIMARY OUTCOMES:
Overall survival defines as the time between the date of surgery and death or date of last news | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France